CLINICAL TRIAL: NCT01504295
Title: A Novel Pharmacotherapy for Alcoholism and Alcohol Liver Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, George Kenna, Assistant Professor of Psychiatry, Brown University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AA021128; R21AA021128 (NIH)
Record Dates: First submitted 2012-01-04; First posted 2012-01-05 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Alcoholism,; Alcoholic Liver Disease
MeSH Terms: conditions — Alcoholism; Liver Diseases, Alcoholic | interventions — metadoxine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metadoxine (Experimental): Metadoxine 500mg tablet t.i.d.for 12 weeks
  Interventions: Drug: Metadoxine
- Sugar pill (Placebo Comparator): Placebo group
  Interventions: Drug: Metadoxine

INTERVENTIONS:
Drug: Metadoxine — Improve Liver Function and Reduce ALcohol Use

SUMMARY:
It is proposed to test metadoxine (MTDX) that it is hypothesized to be significantly beneficial for the treatment of alcoholism and ALD. Metadoxine is currently approved in Europe for acute and chronic alcohol intoxication but has never been tested in the US. Furthermore, MTDX is used in Europe to treat ALD. Preliminary evidence shows that MTDX reduces alcohol consumption in AD individuals. If the role of MTDX in reducing alcohol consumption and improve liver function is confirmed by a rigorous study design, then MTDX might represent a truly innovative pharmacotherapy for AD, given the potential to be used for AD individuals with ALD. However until this proposal, MTDX has never been investigated as a treatment for AD able to reduce both alcohol consumption and improve alcohol-related liver damage via a double-blind placebo-controlled study. This project therefore proposes to conduct a 12-week (followed by a 3-month follow-up), double-blind, placebo-controlled, between-subject randomized clinical trial with MTDX (500mg t.i.d.) in AD individuals.

DETAILED DESCRIPTION:
Treatments for ALD have limited success when drinking continues. Cessation of alcohol consumption or a significant reduction in alcohol intake improves histology and survival of patients with any stage of ALD. While alcohol abstinence may not be sufficient to provide a total recovery of ALD, patients with uncomplicated ALD have a 5-year survival of almost 90% if they stop drinking. Consequently, abstinence is the most important therapeutic intervention for patients with ALD. When combined with psychosocial treatments, currently approved medications can improve outcomes for some AD individuals; however, these treatments are unsuccessful for many others. One of the limiting factors that must be taken into consideration when using currently approved medications such as disulfiram or naltrexone is liver function. Given their hepatic metabolism, disulfiram or naltrexone both increase the risk of hepatotoxicity in AD individuals. Therefore, a pharmacotherapy that is effective for AD, that is safe for the liver and able to recover alcohol-related liver damage thereby improving liver function, would be an ideal medication. However as of now, no drug has been found to provide all of these benefits to AD individuals. It is proposed therefore to test metadoxine (MTDX) that it is hypothesized is significantly beneficial for the treatment of alcoholism and ALD. Metadoxine is currently approved in Europe for acute and chronic alcohol intoxication but has never been tested in the US. Furthermore, MTDX is used in Europe to treat ALD. Preliminary evidence shows that MTDX reduces alcohol consumption in AD individuals. If the role of MTDX in reducing alcohol consumption and improve liver function is confirmed by a rigorous study design, then MTDX might represent a truly innovative pharmacotherapy for AD, given the potential to be used for AD individuals with ALD. However until this proposal, MTDX has never been investigated as a treatment for AD able to reduce both alcohol consumption and improve alcohol-related liver damage via a double-blind placebo-controlled study. This project therefore proposes to conduct a 12-week (followed by a 3-month follow-up), double-blind, placebo-controlled, between-subject randomized clinical trial with MTDX (500mg t.i.d.) in AD individuals.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18;
* females must be post-menopausal for ≥1 year, surgically sterile, or practicing a birth control before entry and throughout the study; have a negative urine pregnancy test at screening and before randomization;
* current DSM-IV diagnosis of alcohol use disorder (or if relevant at study start-DSM-V) with current (i.e. past 90 days prior to screening) "at-risk" drinking defined as an average overall consumption of ≥28 drinks/week for men and ≥21 drinks/week for women;
* desire abstinence;
* evidence of alcoholic liver disease (ALD) based on a thorough history, physical examination, and laboratory tests (i.e. the De Ritis ratio of AST:ALT ratio ~2:1), which is characteristic of ALD.

Exclusion Criteria:

* lifetime DSM diagnosis of schizophrenia, bipolar disorder, or other psychosis;
* in the investigators' opinion, risk of suicide (e.g. active plan, or recent attempt in last year);
* current DSM-IV diagnosis of dependence on any psychoactive substance other than alcohol and nicotine;
* repeated positive urine screen for any substance other than marijuana;
* history of hospitalization for alcohol intoxication delirium or alcohol withdrawal delirium;
* Clinical Institute Withdrawal Assessment for Alcohol (CIWA-Ar) score >10, at any assessment;
* having received a psychological and/or pharmacological treatment for alcohol or having participated in a treatment research study within the past 90 days;
* having participated in any clinical trial with an investigational agent within the past 30 days;
* treatment with levodopa/carbidopa or reported diagnosis of Parkinson's disease;
* AST and/or ALT >10 x upper normal limit; Child-Pugh-Turcotte (CPT) score stage C, model for end-stage liver disease (MELD) score >21 (CPT and MELD scores are assessed by blood tests - e.g. bilirubin, albumin, INR, Cr - and medical history); and/or medical history positive for decompensated liver disease (ascites, encephalopathy, variceal bleeding or hepatorenal syndrome) and/or medical history positive for hepatocellular carcinoma; 11) history of allergy to MTDX or PCA and pyridoxol;
* other serious illnesses, e.g. kidney failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-04; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Percent Days Abstinent (PDA) | 12 weeks
  We hypothesize that metadoxine (MTDX), compared to placebo significantly increases percent days abstinent (PDA) during the 12 weeks of drug administration, as measured by the timeline follow-back (TLFB).

SECONDARY OUTCOMES:
Follow-up PDA | 12 weeks
  We hypothesize that MTDX, compared to placebo results in significantly higher PDA from discontinuation of the medication to the 3-month follow-up, as measured by the TLFB.
Adverse Events | 12 weeks
  We hypothesize that MTDX, compared to placebo has no greater frequency and intensity of Adverse Events (AE).

CONTACTS AND LOCATIONS:
Overall Officials: George A Kenna, PhD RPh, Principal Investigator — Brown University
Locations (1):
- Brown University Center for Alcohol and Addiction Studies, Providence, Rhode Island, United States

REFERENCES:
- [Background] Shpilenya LS, Muzychenko AP, Gasbarrini G, Addolorato G. Metadoxine in acute alcohol intoxication: a double-blind, randomized, placebo-controlled study. Alcohol Clin Exp Res. 2002 Mar;26(3):340-6. PMID 11923586
- [Background] Addolorato G, Ancona C, Capristo E, Gasbarrini G. Metadoxine in the treatment of acute and chronic alcoholism: a review. Int J Immunopathol Pharmacol. 2003 Sep-Dec;16(3):207-14. doi: 10.1177/039463200301600304. PMID 14611722
- [Background] Leggio L, Kenna GA, Ferrulli A, Zywiak WH, Caputo F, Swift RM, Addolorato G. Preliminary findings on the use of metadoxine for the treatment of alcohol dependence and alcoholic liver disease. Hum Psychopharmacol. 2011 Dec;26(8):554-9. doi: 10.1002/hup.1244. Epub 2011 Nov 16. PMID 22095793
- [Background] Guerrini I, Gentili C, Nelli G, Guazzelli M. A follow up study on the efficacy of metadoxine in the treatment of alcohol dependence. Subst Abuse Treat Prev Policy. 2006 Dec 18;1:35. doi: 10.1186/1747-597X-1-35. PMID 17176456
- [Background] Caballeria J, Pares A, Bru C, Mercader J, Garcia Plaza A, Caballeria L, Clemente G, Rodrigo L, Rodes J. Metadoxine accelerates fatty liver recovery in alcoholic patients: results of a randomized double-blind, placebo-control trial. Spanish Group for the Study of Alcoholic Fatty Liver. J Hepatol. 1998 Jan;28(1):54-60. doi: 10.1016/s0168-8278(98)80202-x. PMID 9537864